CLINICAL TRIAL: NCT02887053
Title: Développement Méthodologique de l'Imagerie Par Résonance Magnétique (IRM)
Brief Title: Methodological Developments for Magnetic Resonance Imaging (MRI)
Acronym: METHODO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Valérie LAURENT, Principal Investigator, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2008-A01209-46
Record Dates: First submitted 2016-07-15; First posted 2016-09-01 (Estimated); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Healthy Subjects
Keywords: MRI; Healthy subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All subjects (Experimental): All subjects will have an MRI examination
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI

SUMMARY:
The purpose of this study is to optimize clinical MR protocols and to validate MR acquisition parameters.

ELIGIBILITY:
Inclusion Criteria:

* to be over 18 year-old,
* to be able to give an informed consent,
* to have underwent a pre-inclusion medical examination,
* to present no contraindication to MR examination,
* to be enrolled in a social security plan.

Exclusion Criteria:

* subject refusal,
* subject under a measure of legal protection,
* any contraindication to MR examination (active medical device, ferromagnetic foreign body, pregnancy, morbid obesity, claustrophobia, … ).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1807 (Actual)
Dates: Start 2008-11 (Actual); Primary Completion 2022-05-26 (Actual); Study Completion 2022-05-26 (Actual)

PRIMARY OUTCOMES:
Image quality based on standard imaging quality criteria | 6 months after the last inclusion
  Image quality criteria will be :
  * Signal to Noise Ratio and Contrast to Noise Ratio measured in arbitrary units.
  * absence of blurring and artefacts will be assessed by at least one radiologist according to an ordinal scale

SECONDARY OUTCOMES:
T1/T2 Quantitative sub studies | 6 months after the last inclusion
  For quantitative studies such as T1/T2 studies a T1/T2 quantification will be calculated. These parameters will be reported in ms.
Brain Functional MRI sub studies | 6 months after the last inclusion
  For functional MRI studies, brain activity will be described in terms of brain localisation based on blood oxygen level-dependent signal variation and its intensity.
Cardiac function MRI sub studies: volume | 6 months after the last inclusion
  For cardiac imaging, cardiac function will be evaluated. Parameters such as left ventricle (LV) and right ventricle (RV) end-diastolic volumes end-systolic volumes will be measured and reported in mL/m².
Cardiac mass MRI sub studies: mass | 6 months after the last inclusion
  For cardiac imaging, cardiac function will be evaluated. LV and RV mass index will be measured and reported in g/m2.
Cardiac function MRI sub studies: ejection fraction | 6 months after the last inclusion
  For cardiac imaging, cardiac function will be evaluated. Ejection fraction for both ventricles will be calculated and reported in %.
Diffusion weighted MRI sub studies | 6 months after the last inclusion
  For diffusion studies, the apparent diffusion coefficient (ADC) whic is a measure of the magnitude of diffusion (of water molecules) within tissue will be estimated (mm2/s).
Diffusion tensor MRI sub studies | 6 months after the last inclusion
  The fractional anisotropy (FA) which is a scalar value between zero and one, which describes the degree of anisotropy of a diffusion process, could also be estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Laurent, MD,PhD, Principal Investigator — CHRU de Nancy; Jacques Felblinger, MD,PhD, Principal Investigator — CHRU de Nancy
Locations (1):
- CHRU de Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leclere J, Isaieva K, Drouot G, Gillet R, Felblinger J, Vuissoz PA, Dubernard X. Quantifying symmetry in mandibular condyle motion: a real-time MRI approach. J Oral Facial Pain Headache. 2025 Dec;39(4):227-234. doi: 10.22514/jofph.2025.079. Epub 2025 Dec 12. PMID 41436119